CLINICAL TRIAL: NCT01872871
Title: The Efficacy of Paracetamol in Reducing Pain During Ophthalmological Examination for Retinopathy of Prematurity: a Prospective Randomised Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Serdar Beken, M.D., Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.10.4.İSM.4.06.68.49/231; B.10.4.İSM.4.06.68.49 (Registry Identifier: Sami Ulus)
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- local anasthetic drops (Placebo Comparator): topical anaesthetic drop with placebo
  Interventions: Drug: Topical anaesthetic drop with placebo
- Paracetamol (Active Comparator): Topical anaesthetic drop with Paracetamol
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — paracetamol with local anesthetic eye drop versus placebo with local anesthetic eye drops
  Arms: Paracetamol
Drug: Topical anaesthetic drop with placebo
  Arms: local anasthetic drops

SUMMARY:
Retinopathy of prematurity (ROP) is one of the major morbidity among preterm infants. Although, local anesthetics reduce pain to some extent, eye examination still remains as a painful procedure. The investigators aimed to evaluate the effect of oral paracetamol combined with local anesthetics for pain relief during ophthalmological examination.

ELIGIBILITY:
Inclusion Criteria:

* gestational age below 32 weeks or birth weight below 1500 grams

Exclusion Criteria:

* congenital anomalies, necrotising enterocolitis, surgical problems

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-08 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Reducing pain assessment score | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sami Ulus Childrens Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Allegaert K, Tibboel D, Naulaers G, Tison D, De Jonge A, Van Dijk M, Vanhole C, Devlieger H. Systematic evaluation of pain in neonates: effect on the number of intravenous analgesics prescribed. Eur J Clin Pharmacol. 2003 Jun;59(2):87-90. doi: 10.1007/s00228-003-0585-3. Epub 2003 Apr 4. PMID 12682806